CLINICAL TRIAL: NCT03889730
Title: Impact of Intraoperative Hypotension on Risk of Acute Kidney Injury After Off-pump Coronary Artery Bypass Grafting Surgery: A Retrospective Cohort Study
Brief Title: Intraoperative Hypotension and Acute Kidney Injury After Off-pump Coronary Artery Bypass Grafting Surgery
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anaesthesiology and Critical Care Medicine, Peking University First Hospital
Other Study IDs: OPCABG-AKI-BP
Record Dates: First submitted 2019-03-23; First posted 2019-03-26 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Coronary Artery Bypass, Off-Pump; Intraoperative Hypotension; Acute Kidney Injury
Keywords: Coronary Artery Bypass, Off-Pump; Intraoperative Hypotension; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute renal injury (AKI) is a common complication after cardiac surgery and is associated with worse outcomes. Hypotension is an important risk factor for the development of AKI after noncardiac surgery. However, the association between intraoperative hypotension and AKI after cardiac surgery has not been fully investigated. The purpose of this study is to analyze the association between intraoperative hypotension and acute kidney injury after off-pump coronary artery bypass surgery.

DETAILED DESCRIPTION:
Acute renal injury (AKI) is a common complication after cardiac surgery. Cardiac surgery-associated acute kidney injury (CSA-AKI) is associated with increased in-hospital mortality, prolonged length of stay in the Intensive Care Unit and hospital, and higher costs of care. Intraoperative hypotension is an important risk factor for the development of AKI after noncardiac surgery. In a retrospective analysis, a mean arterial pressure of less than 55 mmHg predicted the occurrence of adverse cardiac- and renal-related outcomes after noncardiac surgery. Other studies also revealed that intraoperative hypotension is associated with increased incidence of AKI and 1-year mortality after noncardiac surgery. In patients undergoing cardiac surgery, 30-day mortality is proportionate to the extent of systolic blood pressure excursions outside the range of 75 to 135 mm Hg intraoperatively. However, the correlation between intraoperative hypotension and the development of AKI after cardiac surgery has not been fully investigated. The purpose of this study is to analyze the association between intraoperative hypotension and the risk of acute kidney injury after off-pump coronary artery bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years;
* Underwent off-pump CABG surgery.

Exclusion Criteria:

* End-stage renal disease requiring renal-replacement therapy;
* Emergency surgery;
* Kidney transplantation within 3 months;
* Missing data.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing off-pump coronry artery bypass grafting surgery from April 2012 to March 2018 in Peking University First Hospital
Sampling Method: Non-Probability Sample
Enrollment: 821 (Actual)
Dates: Start 2019-03-03 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Incidence of acute kidney injury (AKI) within 7 days after surgery | Up to 7 days after surgery
  Development of AKI within 7 days after surgery is diagnosed according to the Kidney Disease Improving Global Outcomes (KDIGO) criteria

SECONDARY OUTCOMES:
Classification of AKI within 7 days after surgery | Up to 7 days after surgery
  Development of AKI within 7 days after surgery is diagnosed according to the KDIGO criteria
Duration of mechanical ventilation after surgery | Up to 30 days after surgery
  Duration of mechanical ventilation after surgery
Length of stay in hospital after surgery | Up to 30 days after surgery
  Length of stay in hospital after surgery
Length of stay in intensive care unit (ICU) after surgery | Up to 30 days after surgery
  Length of stay in intensive care unit (ICU) after surgery
Incidence of major adverse cardiovascular events (MACEs) within 30 days after surgery | Up to 30 days after surgery
  MACEs within 30 days after surgery include cardiovascular death, non-fatal cardiac arrest, acute myocardial infarction, revascularization, and ischemic stroke.
Incidence of non-MACE complications within 30 days after surgery | Up to 30 days after surgery
  Non-MACE complications within 30 days after surgery indicate new-onset medical conditions other than MACEs that produce harmful effects on patients' recovery and required therapeutic intervention.
All-cause mortality in hospital | Up to 30 days after surgery
  All-cause mortality in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bove T, Monaco F, Covello RD, Zangrillo A. Acute renal failure and cardiac surgery. HSR Proc Intensive Care Cardiovasc Anesth. 2009;1(3):13-21. PMID 23439962
- [Background] Hobson CE, Yavas S, Segal MS, Schold JD, Tribble CG, Layon AJ, Bihorac A. Acute kidney injury is associated with increased long-term mortality after cardiothoracic surgery. Circulation. 2009 May 12;119(18):2444-53. doi: 10.1161/CIRCULATIONAHA.108.800011. Epub 2009 Apr 27. PMID 19398670
- [Background] Ortega-Loubon C, Fernandez-Molina M, Carrascal-Hinojal Y, Fulquet-Carreras E. Cardiac surgery-associated acute kidney injury. Ann Card Anaesth. 2016 Oct-Dec;19(4):687-698. doi: 10.4103/0971-9784.191578. PMID 27716701
- [Background] Coleman MD, Shaefi S, Sladen RN. Preventing acute kidney injury after cardiac surgery. Curr Opin Anaesthesiol. 2011 Feb;24(1):70-6. doi: 10.1097/ACO.0b013e3283422ebc. PMID 21157303
- [Background] Sun LY, Wijeysundera DN, Tait GA, Beattie WS. Association of intraoperative hypotension with acute kidney injury after elective noncardiac surgery. Anesthesiology. 2015 Sep;123(3):515-23. doi: 10.1097/ALN.0000000000000765. PMID 26181335
- [Background] Abbott TEF, Pearse RM, Archbold RA, Ahmad T, Niebrzegowska E, Wragg A, Rodseth RN, Devereaux PJ, Ackland GL. A Prospective International Multicentre Cohort Study of Intraoperative Heart Rate and Systolic Blood Pressure and Myocardial Injury After Noncardiac Surgery: Results of the VISION Study. Anesth Analg. 2018 Jun;126(6):1936-1945. doi: 10.1213/ANE.0000000000002560. PMID 29077608
- [Background] Aronson S, Dyke CM, Levy JH, Cheung AT, Lumb PD, Avery EG, Hu MY, Newman MF. Does perioperative systolic blood pressure variability predict mortality after cardiac surgery? An exploratory analysis of the ECLIPSE trials. Anesth Analg. 2011 Jul;113(1):19-30. doi: 10.1213/ANE.0b013e31820f9231. Epub 2011 Feb 23. PMID 21346163
- [Background] Bijker JB, van Klei WA, Vergouwe Y, Eleveld DJ, van Wolfswinkel L, Moons KG, Kalkman CJ. Intraoperative hypotension and 1-year mortality after noncardiac surgery. Anesthesiology. 2009 Dec;111(6):1217-26. doi: 10.1097/ALN.0b013e3181c14930. PMID 19934864
- [Background] Schopka S, Diez C, Camboni D, Floerchinger B, Schmid C, Hilker M. Impact of cardiopulmonary bypass on acute kidney injury following coronary artery bypass grafting: a matched pair analysis. J Cardiothorac Surg. 2014 Jan 18;9:20. doi: 10.1186/1749-8090-9-20. PMID 24438155
- [Background] Rosner MH, Okusa MD. Acute kidney injury associated with cardiac surgery. Clin J Am Soc Nephrol. 2006 Jan;1(1):19-32. doi: 10.2215/CJN.00240605. Epub 2005 Oct 19. PMID 17699187
- [Background] Kheterpal S, Tremper KK, Heung M, Rosenberg AL, Englesbe M, Shanks AM, Campbell DA Jr. Development and validation of an acute kidney injury risk index for patients undergoing general surgery: results from a national data set. Anesthesiology. 2009 Mar;110(3):505-15. doi: 10.1097/ALN.0b013e3181979440. PMID 19212261
- [Background] Kellum JA, Lameire N; KDIGO AKI Guideline Work Group. Diagnosis, evaluation, and management of acute kidney injury: a KDIGO summary (Part 1). Crit Care. 2013 Feb 4;17(1):204. doi: 10.1186/cc11454. PMID 23394211